CLINICAL TRIAL: NCT01084967
Title: Study of Clinical Characteristics and Genetic Susceptibility in Chinese Obese Youngs
Brief Title: Genetics of Obesity in Chinese Youngs
Acronym: GOCY
Status: Recruiting | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Guang Ning, Director, Shanghai Jiao Tong University School of Medicine
Other Study IDs: CCEMD008
Record Dates: First submitted 2010-03-10; First posted 2010-03-11 (Estimated); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Obesity; Metabolic Syndrome
Keywords: obesity; metabolic syndrome; genetic risk markers; copy number variation
MeSH Terms: conditions — Obesity; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood,fasting serum, morning urine and feces
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy lean control group: The healthy lean controls consisted of age-, sex- and geography-matched young volunteers, or "golden standard" lean controls from China Cardiometabolic Disease and Cancer Cohort Study (4C Study).
  Healthy volunteers:
  1. BMI:18.5-22.9kg/m2;
  2. Age:14-30 years old;
  3. To be proved normal by the examinations of liver and kidney function,blood lipids profile,FBG, PBG, fasting insulin and HbA1c.
  Controls from 4C Study:
  1. 17.0≤BMI≤23.0kg/m2 and waist circumference <85cm for males and <80cm for females;
  2. 1.8≤LDL-c≤3.4mmol/l;
  3. FBG<6.1, PBG<7.8;
  4. HOMA-IR<2.5;
  5. BP <140/90mmHg;
  6. eGFR>60mL/(min·1.73 m2), ALT<40IU/L, AST<40IU/L;
  7. Excluding the history of hyperthyroidism, digestive system diseases, malignant tumors, infectious diseases (hepatitis B) and other systemic wasting diseases; Severe dysfunction of heart, lung and kidney;
  8. Not using antihypertensive, hypoglycemic and lipid-lowering drugs；
  9. No history of smoking.
- obesity group: 1. BMI ≥30kg/m2;
  2. Age:14-30 years old; obesity group 4000, lean healthy control group 4000

SUMMARY:
The purpose of this study is to explore the pathogenesis and genetic susceptibility of obese subjects,providing a convincing argument for further treatment of obesity and metabolic syndrome.

DETAILED DESCRIPTION:
Obesity has become a major worldwide challenge to public health, owing to an interaction between the obesogenic environment and a strong genetic contribution.Previous studies found that genetic factors determine 40%-70% of obese phenotype.Under such circumstances, the screening of obesity susceptibility gene is particularly important for society or family to take measures to prevent obesity.

Recent extensive genome-wide association studies(GWASs) have identified numerous single nucleotide polymorphisms associated with obesity,but these loci together account for only a small fraction of the known heritable component.Two studies in 2010 Nature,for the first time, put rare copy number variation (CNV)in association with severe early-onset obesity.Their significance lie not only in the discovery of the pathogenic genes of severe early-onset obesity but,more importantly,in providing new strategies for finding out genes that cause complex diseases.

Obese patients and healthy lean controls proved by a series of blood biochemical examinations will be enrolled in this study.The present study intends to use the techniques such as enzyme-linked immunosorbent assay, real-time fluorescence quantitative PCR,gene chip,construction of viral vectors,transfection, taking advantage of the established database,by means of serum assays and functional tests, associate copy number variation with obesity phenotype to explain the root cause of obesity.Meanwhile biomarkers, gut flora and genetic risk factors will be evaluated in the study subjects.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI)≥ 30kg/m2
* predominantly east China to minimize population stratification
* willing and able to provide informed consent

Exclusion Criteria:

* pregnancy/lactation
* Cushing syndrome
* Hypothyroidism
* obesity caused by pituitary and hypothalamic lesions
* drug related obesity
* history of major psychiatric illness

Ages: 14 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The population from which cohorts will be selected include students, residents, staff, and/or faculty who are present on Shanghai Jiaotong University school of medicine, and surrounding areas.
Sampling Method: Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2009-03; Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Guang Ning, MD.PhD, Study Chair — Shanghai Jiao Tong University School of Medicine; Jie Hong, MD, Principal Investigator — Shanghai Jiao Tong University School of Medicine; Jiqiu Wang, MD.PhD, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Hong J, Bo T, Xi L, Xu X, He N, Zhan Y, Li W, Liang P, Chen Y, Shi J, Li D, Yan F, Gu W, Wang W, Liu R, Wang J, Wang Z, Ning G. Reversal of Functional Brain Activity Related to Gut Microbiome and Hormones After VSG Surgery in Patients With Obesity. J Clin Endocrinol Metab. 2021 Aug 18;106(9):e3619-e3633. doi: 10.1210/clinem/dgab297. PMID 33950216